CLINICAL TRIAL: NCT03133234
Title: An Observational, Retrospective, Real World Study of Osimertinib in Ethnic Chinese Patients With Locally Advanced/Metastatic T790M Mutation-Positive Non-small-cell Lung Cancer (NSCLC )Progressed on Previous Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor (TKI).
Brief Title: Effect of Osimertinib in Ethnic Chinese With EGFR and T790M Mutated NSCLC
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5160R00016
Record Dates: First submitted 2017-04-13; First posted 2017-04-28 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: T790M Positive NSCLC Patients
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- EGFR T790M Patients: Patients with locally advanced/metastatic EGFR T790M positive NSCLC progressed on previous EGFR TKI
  Interventions: Drug: osimertinib

INTERVENTIONS:
Drug: osimertinib — Oral dose of 80mg once daily

SUMMARY:
To assess the effectiveness and safety of osimertinib treatment in a real world setting.

DETAILED DESCRIPTION:
The current study will not only assess the effectiveness of osimertinib treatment in a real world setting, but will also help us to understand the real-world testing patterns among T790M mutation positive locally advanced or metastatic NSCLC patients who have progressed after EGFR TKI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age;
* Locally advanced (stage IIIB) or metastatic (stage IV) NSCLC, not amenable to curative surgery or radiotherapy
* Confirmed T790M mutation
* Progressed on previous EGFR TKI treatment. Patients may have also received additional lines of treatment
* Received osimertinib treatment in the participating site between May 1st and Oct 31st 2016

Exclusion Criteria:

• Enrolment in studies that prohibit any participation in this observational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced or metastatic T790M mutation-positive NSCLC patients progressed after EGFR TKI treatment.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
ORR | Followed up with 6 months after last patient in
  Overall response rate (ORR), defined as the proportion of patients with a best response of "responding" to treatment by investigator assessment

SECONDARY OUTCOMES:
PFS | Followed up 10 months after last subject in
  Progression free survival (PFS), defined as the time from the date of first dose of osimertinib to the date of investigator-assessed disease progression or death from any cause during study. Subjects who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment
T790M mutation testing time | Within 14 days after enrollment date
  Average turnaround time.
Treatment patterns | Followed up 10 months after last patient in
  To assess by number of previous adopted/current/future therapies as recorded on the case report form
Adverse events | Follow up 10 months after last patient in.
  To assess by number of adverse events as recorded on the case report form.
Adverse event intensity | Follow up 10 months after last patient in.
  To assess by intensity of adverse events as recorded on the case report form, which will be measured by CTCAE grade system
T790M mutation testing sample | Within 14 days after enrollment date
  To assess by proportion of testing samples types as recorded on the case report form.
T790M mutation testing platform | Within 14 days after enrollment date
  To assess by proportion of each testing platform as recorded on the case report form.
EGFR testing mutation subtype | Within 14 days after enrollment date
  To assess by proportion of EGFR mutation subtype as recorded on the case report form

CONTACTS AND LOCATIONS:
Overall Officials: Yabing Cao, Principal Investigator — Kiang Wu Hospital
Locations (1):
- Kiang Wu Hospital, Macau, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao Y, Qiu X, Xiao G, Hu H, Lin T. Effectiveness and safety of osimertinib in patients with metastatic EGFR T790M-positive NSCLC: An observational real-world study. PLoS One. 2019 Aug 23;14(8):e0221575. doi: 10.1371/journal.pone.0221575. eCollection 2019. PMID 31442277
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14680&filename=Study%20report%20%20of%20osimertinib%20retrospective%20RWE%20study%20in%20Macau.pdf